CLINICAL TRIAL: NCT01719705
Title: Efficacy of Preoperative Pregabalin on the Post-caesarean Pain; a Dose-response Study
Brief Title: Effects of Pregabalin on Post-cesarean Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed R El Tahan, Associate Professor of Anesthesiology & SICU, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R/60
Record Dates: First submitted 2012-10-28; First posted 2012-11-01 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Uncomplicated Singleton Pregnancies
Keywords: caesarean delivery; spinal anesthesia; pregabalin; postoperative pain; morphine
MeSH Terms: conditions — Pain, Postoperative | interventions — Pregabalin; Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): receive two identical placebo capsules
  Interventions: Drug: Placebo
- Pregabalin 150 mg group (Active Comparator): one capsule of pregabalin 150 mg
  Interventions: Drug: Pregabalin 150 mg group
- Pregabalin 300 mg group (Active Comparator): two capsules of pregabalin 150 mg
  Interventions: Drug: Pregabalin 300 mg group

INTERVENTIONS:
Drug: Placebo — Ninety minutes before surgery, the parturients receive two identical placebo capsules
  Arms: Placebo
Drug: Pregabalin 300 mg group — Ninety minutes before surgery, the parturients receive two capsules of pregabalin 150 mg
  Arms: Pregabalin 300 mg group
Drug: Pregabalin 150 mg group — Ninety minutes before surgery, the parturients receive one capsule of pregabalin 150 mg and one placebo capsule
  Arms: Pregabalin 150 mg group

SUMMARY:
Post-cesarean pain management is essential for early mobilization of the mother so that she becomes able to care of her newborn. There choices for postoperative analgesia include spinal, systemic, or both opioids, non-steroidal anti-inflammatory drugs (NSAIDs), local anesthetic infiltrations of the wound, or transverse abdominis plane blocks, which are determined by drug availability, regional and individual preferences, resource limitations and financial considerations. The use of opioids is associated with adverse effects such as nausea, pruritus, sedation, and occasionally respiratory depression.

Pregabalin is an anticonvulsant drug structurally related to the inhibitory neurotransmitter gamma amino butyric acid, that exerts its action by binding to the α-2-δ subunit of the voltage-dependent calcium channel. It reduces the release of the excitatory neurotransmitters and inhibits the hyperalgesia and central sensitization.

A recent meta-analysis demonstrated that pregabalin reduce the postoperative 24 hours cumulative opioid consumption and opioid-related adverse effects namely, vomiting and visual disturbances after surgery. Compared with the use of pregabalin doses lower than 300 mg, the use of doses higher than 300 mg even reduced opioid consumption by 35%.

It is not known if pregabalin is excreted in human milk. There is a case report on the extensive excretion of pregabalin in breast milk, but with low measured concentrations in infant as a consequence of maternal exposure during breast feeding. Food and Drug Administration recommends to discontinue nursing or to discontinue pregabalin in nursing mothers. Pre-delivery single exposure to pregabalin is expected to be safe for the newborns.

Up to the authors' best knowledge, this is the first clinical study on the efficacy and safety of the administration of pregabalin before cesarean delivery.

We hypothesis that the preoperative administration of a single dose of pregabalin will improve the quality of postoperative analgesia after cesarean delivery.

This placebo-controlled study aims to compare the effects of preoperative administrations of single oral doses of pregabalin 150 mg and 300 mg on the postoperative pain scores, cumulative patient controlled morphine consumptions, neonatal Apgar and neurologic and adaptive capacity scores (NACS), and maternal and neonatal adverse effects in parturients scheduled to elective Cesarean delivery under spinal anesthesia.

DETAILED DESCRIPTION:
An independent investigator who will not be involved in the study will instruct the patients preoperatively about the use of patient controlled analgesia and visual analogue scale to assess the severity of postoperative pain (0 mm for no pain and100 mm for worst imaginable pain).

Anaesthetic management will be standardized. Oral ranitidine 150 mg and metoclopramide 10 mg will be given the night before and on the morning of surgery, with 0.3 mol/L sodium citrate 30 mL given 15 min before induction.

Ninety minutes before surgery, subjects will be allocated randomly into three groups by drawing sequentially numbered sealed opaque envelopes containing a software-generated randomization code to the placebo (n = 45), pregabalin 150 mg (n = 45) and the pregabalin 300 mg (n = 45) groups. The placebo and pregabalin capsules look identical and will be prepared by a local pharmacy. An anaesthesiologist not otherwise involved in the study and who will be blinded to treatment regimen will provide perioperative care. An independent investigator will collect perioperative data. All staff in the operating room will be unaware of patient allocation group.

Maternal monitoring will include electrocardiography, non-invasive blood pressure, and pulse oximetry. Left uterine displacement will be maintained.

Spinal anesthesia will be performed in all cases in sitting position at L3-L4 or L4-L5 spaces with hyperbaric bupivacaine 0.5% (12.5 mg) and fentanyl 20 µg. After the umbilical cord is clamped, a 10 IU infusion of oxytocin in 500 mL of lactated Ringer's solution will be infused.

A paediatrician blinded to study group allocation will record Apgar scores at 1 and 5 min, umbilical cord blood gas analysis and NACS at 15 min, 2h, 24 and 48 h after delivery. NACS gives a maximum of 40 with a score >35 denoting vigor.The percentage of infants scoring <35 will be determined.

Postoperative analgesic regime will be standardized in all patients with 12-hourly intramuscular diclofenac 75 mg started immediately at the end of surgery and morphine via patient-controlled analgesia (PCA): 1 mg bolus with an 8 minutes lockout. Postoperative nausea or vomiting will be treated with intravenous metoclopramide 10 mg as required.

Statistical analysis:

Based on a previous study,7 the mean postoperative cumulative morphine consumption at 24 h after caesarean delivery was 38 mg with a standard deviation of 14 mg. An a priori power analysis indicated that 45 subjects were required in each group to detect a 25% reduction in the cumulative morphine consumption at 24 h after caesarean delivery, that was assumed to have a clinically significant effect, with a type-I error of 0.0167 (0.05/3 possible comparisons) and a power of 90%. Additional patients (10%) were included for a final sample size of 150 patients to account for patient dropout during the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* spinal anesthesia
* elective cesarean delivery
* breech presentation
* cephalopelvic disproportion
* previous caesarean delivery
* American Society of Anesthesiologists class I and II

Exclusion Criteria:

* communication barriers
* cardiovascular diseases
* renal diseases
* hepatic diseases
* endocrinal diseases
* neuropsychiatric diseases
* morbid obesity
* diabetes mellitus
* anaemia
* bleeding disorders
* prolonged P-R interval
* hypersensitivity to pregabalin
* receiving pregabalin
* receiving anticonvulsants
* receiving antidepressants
* receiving antipsychotics
* alcohol or drug abuse
* Opiates abuse
* benzodiazepines during the last week
* pregnancy-induced hypertension
* evidence of intrauterine growth restriction
* fetal compromise

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 135 (Actual)
Dates: Start 2012-11; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
cumulative patient controlled morphine consumptions | 24 hours after delivery
  cumulative patient controlled morphine consumptions 24 hours after delivery

SECONDARY OUTCOMES:
postoperative pain scores | 1, 4, 6, 12, 24 and 48 hours after delivery
  visual analogue scale to assess the severity of postoperative pain (0 mm for no pain and100 mm for worst imaginable pain) at rest and on movement
neonatal Apgar scores | 1 and 5 min aftr delivery
Neurologic and adaptive capacity scores | at 15 min, 2h, 24 and 48 h after delivery
  NACS gives a maximum of 40 with a score >35 denoting vigor.The percentage of infants scoring <35 will be determined.
Maternal sedation | every two hours after delivery, for 48 hours after delivery
  sedation (0, alert; 1, somnolent easy to arouse; 2, somnolent difficult to arouse or asleep; 3, not arousable)
Maternal nausea and vomiting | at 24 hours after delivery
  nausea and vomiting (0: no nausea; 1: nausea no vomiting; 2: nausea and vomiting),

OTHER OUTCOMES:
Adverse effects | 24 hours after delivery
  difficulties in lactation, pruritus, dry mouth, flatulence, hypoglycaemia, dizziness, somnolence, ataxia, vertigo, confusion, incoordination, tremor, dyspnoea, blurred or abnormal vision

CONTACTS AND LOCATIONS:
Overall Officials: Samah A El Kenany, MD, Principal Investigator — Anethesiology Dept, College of Medicine, Mansoura University; Mohamed R El Tahan, M.D., Study Chair — Mansoura University
Locations (2):
- Egypt (2):
  - College of Medicine, Mansoura University, Al Mansurah, DK
  - Mansoura University Hospitals, Al Mansurah, DK